CLINICAL TRIAL: NCT07139964
Title: Effectiveness of High-Dose Vitamin D3 in Improving Diabetic Foot Ulcer Healing by Reducing the MMP-9 to TIMP-1 Ratio: Randomized Double-Blind Placebo-Controlled Trial
Brief Title: High-Dose Vitamin D3 for Diabetic Foot Ulcer Healing: Randomized Controlled Trial
Acronym: DFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DP.04.03/D.XVIII.6.8/ETIK/106/
Record Dates: First submitted 2025-08-15; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer; Vitamin D Deficiency; Wound Healing Disorder
Keywords: Diabetic foot ulcer; Vitamin D3 supplementation
MeSH Terms: conditions — Diabetic Foot; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: High-dose Vitamin D3 (Experimental): Description: Participants receive oral vitamin D3, 10,000 IU daily for 28 days, plus standard care for diabetic foot ulcers.
  Intervention Name: Vitamin D3 (Cholecalciferol) Type: Dietary Supplement Dosage: 10,000 IU daily Duration: 28 days
  Interventions: Dietary Supplement: Vitamin D3
- Placebo Comparator: Placebo (Placebo Comparator): Description: Participants receive oral placebo daily for 28 days, plus standard care for diabetic foot ulcers.
  Intervention Name: Placebo Type: Inactive substance Dosage: Matched placebo daily Duration: 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Participants receive oral vitamin D3 (cholecalciferol) 10,000 IU daily for 28 consecutive days, in addition to standard diabetic foot ulcer care according to hospital protocols. Vitamin D3 is provided in identical-appearing capsules. Compliance is monitored using the MMAS-8 adherence scale.
  Other Names: Cholecalciferol
  Arms: Experimental: High-dose Vitamin D3
Other: Placebo — Participants receive an oral placebo capsule daily for 28 consecutive days, in addition to standard diabetic foot ulcer care according to hospital protocols. The placebo is identical in appearance to the vitamin D3 capsule. Compliance is monitored using the MMAS-8 adherence scale.
  Other Names: Inert capsule
  Arms: Placebo Comparator: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the effectiveness of high-dose vitamin D3 supplementation in improving diabetic foot ulcer (DFU) healing. DFUs are common, serious complications of diabetes, often associated with delayed wound healing due to persistent inflammation, impaired angiogenesis, and imbalances between matrix metalloproteinase-9 (MMP-9) and its tissue inhibitor (TIMP-1). Vitamin D deficiency is prevalent among DFU patients and is linked to impaired fibroblast function, poor angiogenesis, and increased inflammation.

Participants with DFUs and serum vitamin D levels <30 ng/mL will be randomized to receive either 10,000 IU oral vitamin D3 daily or placebo for 28 days, in addition to standard DFU care. Primary outcomes include changes in tissue MMP-9/TIMP-1 expression ratio and wound healing progression. The study will provide evidence on whether high-dose vitamin D3 can serve as a safe, effective adjunctive therapy in DFU management.

DETAILED DESCRIPTION:
Diabetic foot ulcers are a prevalent and serious complication of uncontrolled diabetes, with a significant proportion leading to infection, amputation, and mortality. Delayed wound healing in DFUs is often driven by prolonged inflammation, persistent infection, impaired angiogenesis, and an imbalance between extracellular matrix (ECM) degradation by MMP-9 and inhibition by TIMP-1. Elevated MMP-9 levels disrupt keratinocyte migration, collagen deposition, and epithelial regeneration, while reduced TIMP-1 further compromises healing.

Vitamin D plays a regulatory role in immune modulation, inflammation control, fibroblast activity, and angiogenesis. Observational and interventional studies have shown that vitamin D deficiency is common in DFU patients and is associated with slower healing. Supplementation has been linked to improved wound healing, reduced inflammatory markers, and better microcirculation. Vitamin D may also modulate MMP-9 and TIMP-1 expression, thereby restoring ECM balance.

This study is a double-blind, placebo-controlled, randomized controlled trial conducted at Dr. Mohammad Hoesin General Hospital, Palembang. Eligible participants are adults with DFUs, low serum vitamin D (<30 ng/mL), and no exclusion criteria such as advanced kidney disease, severe liver disease, osteomyelitis, or sepsis. Participants will be randomized into two groups:

Intervention group: Oral vitamin D3, 10,000 IU daily for 28 days Control group: Placebo daily for 28 days Both groups will receive standard DFU care. Compliance will be monitored with the MMAS-8 scale. Primary outcomes are changes in tissue MMP-9 and TIMP-1 expression (assessed by immunohistochemistry) and wound healing parameters. Secondary outcomes include changes in serum vitamin D levels and correlation between vitamin D status and wound healing outcomes.

The study aims to determine whether high-dose vitamin D3 supplementation reduces the MMP-9/TIMP-1 ratio and accelerates wound healing, potentially supporting its use as a standard adjunctive therapy for DFUs.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of diabetic foot ulcer (DFU) Serum 25-hydroxyvitamin D level < 30 ng/mL Willingness and ability to provide written informed consent Ability to comply with study procedures and follow-up visits

Exclusion Criteria:

Currently undergoing cancer treatment Pregnant or breastfeeding Current use of vitamin D supplementation History of autoimmune disease Chronic kidney disease with estimated GFR < 30 mL/min/1.73 m² Abnormal liver function tests (AST or ALT ≥ 3× upper normal limit) Ankle-brachial index (ABI) < 0.4 Presence of osteomyelitis Proven sepsis Allergy to vitamin D3 Amputation prior to randomization Withdrawal of consent during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in tissue MMP-9/TIMP-1 expression ratio from baseline to Day 28 | Baseline (Day 0) and after completion of intervention (Day 28)
  Ratio of matrix metalloproteinase-9 (MMP-9) to tissue inhibitor of metalloproteinase-1 (TIMP-1) expression in wound tissue, measured using immunohistochemistry from surgical biopsy samples.

SECONDARY OUTCOMES:
Change in wound size from baseline to Day 28 | Baseline (Day 0) and Day 28
  Measurement of ulcer area using standardized planimetry software from digital photographs.
Change in serum vitamin D3 concentration from baseline to Day 28 | Baseline (Day 0) and Day 28
  Serum 25-hydroxyvitamin D3 level measured by chemiluminescent immunoassay.
Change in tissue MMP-9 expression from baseline to Day 28 | Baseline (Day 0) and Day 28
  Immunohistochemical staining score of matrix metalloproteinase-9 in wound biopsy specimens.
Change in tissue TIMP-1 expression from baseline to Day 28 | Baseline (Day 0) and Day 28
  Immunohistochemical staining score of tissue inhibitor of metalloproteinase-1 in wound biopsy specimens.
Correlation between serum vitamin D3 level and wound healing outcomes | Baseline (Day 0) to Day 28
  Pearson or Spearman correlation between serum 25-hydroxyvitamin D3 concentration and percentage reduction in ulcer size.

CONTACTS AND LOCATIONS:
Overall Officials: Kemas M Dahlan, M.D., Principal Investigator — Consultant Vascular Surgeon, Department of Surgery, Dr. Mohammad Hoesin General Hospital Palembang
Locations (1):
- Dr. Mohammad Hoesin General Hospital, Palembang, South Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shin MH, Lee Y, Kim MK, Lee DH, Chung JH. UV increases skin-derived 1alpha,25-dihydroxyvitamin D3 production, leading to MMP-1 expression by altering the balance of vitamin D and cholesterol synthesis from 7-dehydrocholesterol. J Steroid Biochem Mol Biol. 2019 Dec;195:105449. doi: 10.1016/j.jsbmb.2019.105449. Epub 2019 Aug 27. PMID 31470109
- [Result] Luanraksa S, Jindatanmanusan P, Boonsiri T, Nimmanon T, Chaovanalikit T, Arnutti P. An MMP/TIMP ratio scoring system as a potential predictive marker of diabetic foot ulcer healing. J Wound Care. 2018 Dec 2;27(12):849-855. doi: 10.12968/jowc.2018.27.12.849. PMID 30557113
- [Result] Kim SH, Baek MS, Yoon DS, Park JS, Yoon BW, Oh BS, Park J, Kim HJ. Vitamin D Inhibits Expression and Activity of Matrix Metalloproteinase in Human Lung Fibroblasts (HFL-1) Cells. Tuberc Respir Dis (Seoul). 2014 Aug;77(2):73-80. doi: 10.4046/trd.2014.77.2.73. Epub 2014 Aug 29. PMID 25237378
- [Result] Masood MQ, Khan A, Awan S, Dar F, Naz S, Naureen G, Saghir S, Jabbar A. COMPARISON OF VITAMIN D REPLACEMENT STRATEGIES WITH HIGH-DOSE INTRAMUSCULAR OR ORAL CHOLECALCIFEROL: A PROSPECTIVE INTERVENTION STUDY. Endocr Pract. 2015 Oct;21(10):1125-33. doi: 10.4158/EP15680.OR. Epub 2015 Jul 7. PMID 26151421
- [Result] Razzaghi R, Pourbagheri H, Momen-Heravi M, Bahmani F, Shadi J, Soleimani Z, Asemi Z. The effects of vitamin D supplementation on wound healing and metabolic status in patients with diabetic foot ulcer: A randomized, double-blind, placebo-controlled trial. J Diabetes Complications. 2017 Apr;31(4):766-772. doi: 10.1016/j.jdiacomp.2016.06.017. Epub 2016 Jun 23. PMID 27363929